CLINICAL TRIAL: NCT01111188
Title: Phase I Trial of PD 0332991 Plus Bortezomib in Patients With Relapsed Mantle Cell Lymphoma
Brief Title: Trial of PD 0332991 Plus Bortezomib in Patients With Relapsed Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0903010300
Record Dates: First submitted 2010-04-19; First posted 2010-04-27 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — palbociclib; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- all subjects (Experimental): Subjects will receive PD 0332991 plus bortezomib. The dose of each agent will be dependent on the time point the subject enters the trial.
  Interventions: Drug: PD 0332991; Drug: bortezomib

INTERVENTIONS:
Drug: PD 0332991 — PD 0332991 will be given on Days 1-12 followed by 9 days of non-treatment in a 21-day cycle. Dose will depend on dose escalation schedule.
  (-3a) 50 mg (-3) 50 mg (-2)75 mg (-1)75 mg (1)100 mg (2)125 mg (3)125 mg (3a)100 mg
  Other Names: Palbociclib
Drug: bortezomib — Given as intravenous bolus on days 8, 11, 15, and 18 of 21-day cycle. Dose depends on dose-escalation schedule.
  (-3a)1.0 mg/m2 (-3) 0.7 mg/m2 (-2) 0.7 mg/m2 (-1) 1.0 mg/m2 ( 1) 1.0 mg/m2 ( 2) 1.0 mg/m2 ( 3) 1.3 mg/m2 (3a)1.3 mg/m2
  Other Names: Velcade

SUMMARY:
Mantle cell lymphoma (MCL) is characterized by cell cycle dysregulation. PD 0332991 is a cyclin-dependent kinase 4 and 6 inhibitor capable of inhibiting cell cycling of MCL. A phase I study has demonstrated the safety and anti-lymphoma activity of PD 0332991. Bortezomib is a first generation proteasome inhibitor approved for treatment of patients with recurrent MCL. Preclinical data suggests that PD 0332991 and bortezomib may act synergistically in MCL.

PD 0332991 will be administered continuously for 12 days followed by a 9 day period without treatment. Bortezomib will be administered by intravenous bolus on days 8, 11, 15, and 18 of each cycle. One cycle is defined as three weeks. A maximum of ten cycles will be administered.

DETAILED DESCRIPTION:
Escalating doses of PD 0332991 in combination with bortezomib will be studied sequentially, with at least 3 patients in each dose level until the MTD is determined. PD 0332991 will be given orally, starting on Day 1 of each cycle, once a day for 12 days followed by 9 days without treatment. Bortezomib will be given by intravenous (IV) bolus or subcutaneously (taking 3 to 5 seconds to administer) on days 8, 11, 15 and 18. For dose levels 3a and 4b, bortezomib will be administered only on days 15 and 18. One cycle is defined as 3 weeks (21 days). Subjects will remain on treatment until they meet criteria for withdrawal from treatment described in section 5.4 (e.g., DLT, disease progression, unacceptable toxicity, or withdrawal of consent).

The pharmacist will maintain records of drug receipt (if applicable), drug preparation, and dispensing, including the applicable lot numbers, patients' height, body weight, and body surface area, and total drug administered in milliliters and milligrams. Any discrepancy between the calculated dose and dose administered and the reason for the discrepancy must be recorded in the source documents.

Treatment will be administered only to eligible patients under the supervision of the investigator or identified sub-investigator (s). Treatment will be administered on an outpatient basis. Reported adverse events and potential risks are described in Section 7. Appropriate dose modifications are described in Section 6. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed mantle cell lymphoma as defined by the World Health Organization. All patients must have either a demonstrated t(11;14) by karyotype, fluorescent in-situ hybridization (FISH) or positive immunohistochemistry for cyclin D1.
* Subjects must have measurable disease, defined as at least one tumor mass of > 1.5 cm in diameter.
* Subjects must have received at least one prior chemotherapy-containing regimen and at least one prior rituximab-containing regimen.
* Age > = 18 years.
* Accessible disease, defined as at least one of the following:

  * Adenopathy accessible to core needle biopsy
  * Bone marrow involvement
  * Circulating lymphoma cells in the peripheral blood
* ECOG performance status < = 2
* Patients must have normal organ and marrow function as defined below within 14 days before enrollment:

  * ANC > = 750 cells/uL
  * platelets > = 75,000 cells/uL
  * Hemoglobin > = 8.0 g/dL
  * total bilirubin < = 1.5 times upper limit of normal
  * AST(SGOT)/ALT(SGPT) < = 3 times upper limit of normal
  * Calculated creatinine clearance > = 30 mL/min
* The effects of bortezomib and PD 0332991 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, female subjects must either be post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) prior to study entry and for the duration of the study. Male subjects must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a female subject become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Subjects must be willing and able to comply with the scheduled visits, treatment plans, laboratory tests, and other procedures

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, antibodies, or investigational agents within 4 weeks prior to entering the study unless progression has been documented while on treatment, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Patients may be receiving prednisone at a maximum dose of 10 mg/day orally, provided the dose has been stable during the prior two weeks before starting treatment.
* Patients may not be receiving any other investigational agents.
* Prior exposure to PD 0332991
* Prior exposure to bortezomib will only be permitted if there was a documented complete or partial response and progression occurred off therapy
* Patients must not have experienced significant hematologic (grade 4) or neuropathic toxicities (grade 3 or 4) due to prior bortezomib therapy
* Peripheral neuropathy > = grade 2 (CTCAEv3.0) within 14 days before enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib (e.g. boron or mannitol).
* Contraindication to serial core needle biopsies
* Known HIV infection
* Known malabsorption syndrome that may affect absorption of the drug
* Known or suspected CNS involvement
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* QTc > 470 msec
* Current use or anticipated need for food or drugs that are known potent CYP3A4 inhibitors, including their administration within 7-days prior to the first PD 0332991dose (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, nefazodone, diltiazem, atazanavir, amprenavir,and fosamprenavir)
* Current use or anticipated need for drugs that are known potent CYP3A4 inducers, including their administration within 14-days prior to the first PD 0332991 dose (i.e. carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, primidone, rifabutin, rifampin, and St. John's Wort).
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 7), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08-23 (Actual); Primary Completion 2013-02-26 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) of PD 0332991 in combination with bortezomib in patients with recurrent mantle cell lymphoma | Days 1-21 of treatment
  MTD will be determined by occurrence of Dose Limiting Toxicities during the first cycle:
  * Any treatment-related grade 3 or 4 non-hematologic toxicity (except alopecia)
  * Delay in the administration of cycle 2 by more than one week due to treatment-related grade 4 neutropenia or thrombocytopenia or treatment-related grade 3-4 non-hematologic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: John P Leonard, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Martin P, Ruan J, Furman R, Rutherford S, Allan J, Chen Z, Huang X, DiLiberto M, Chen-Kiang S, Leonard JP. A phase I trial of palbociclib plus bortezomib in previously treated mantle cell lymphoma. Leuk Lymphoma. 2019 Dec;60(12):2917-2921. doi: 10.1080/10428194.2019.1612062. Epub 2019 May 23. PMID 31120355